CLINICAL TRIAL: NCT02901678
Title: The Effect of Two Different Force Magnitudes on Maxillary Posterior Segment Intrusion in Adult Patients With Skeletal Open Bite Using Temporary Anchorage Devices- A Randomized Clinical Trial
Brief Title: The Effect of Different Force Magnitudes on Maxillary Posterior Segment Intrusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba El-Sayed Kamel Akl, Internal resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 121888
Record Dates: First submitted 2016-09-10; First posted 2016-09-15 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Orthodontics
Keywords: skelatal open bite, posterior intrusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intrusion by 200 g (Active Comparator): Applying 200 g intrusive force for the maxillary posterior segment intrusion using miniscrews
  Interventions: Device: Intrusion by 400 g
- Intrusion by 400 g (Experimental): Applying 400 g of Intrusive force for the maxillary posterior segment intrusion using miniscrews
  Interventions: Device: Intrusion by 400 g

INTERVENTIONS:
Device: Intrusion by 400 g — using miniscrews and coil springs to apply the intrusive force on maxillary posterior segment intrusion.

SUMMARY:
A Randomized clinical trial comparing two different force magnitudes in maxillary posterior segment intrusion in adult patients with skeletal open bite malocclusion

DETAILED DESCRIPTION:
This randomized controlled trial is aiming to study the effect of the different force magnitude on maxillary posterior segment intrusion. Two groups are going to be allocated and the amount and rate of intrusion will be measured and compared.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with an age range from 17 to 25.
* Skeletal open bite.
* Dental open bite that is due to overgrowth of maxillary posterior segment as seen clinically and that can be corrected without surgical intervention (a minimum of 3 mm and a maximum of 8 mm).
* Skeletal class I or mild to moderate skeletal class II that enables camouflage treatment.
* Normal incisor show on smiling (that makes the case indicated for molar intrusion and not for incisor extrusion).
* Full set of maxillary posterior dentition (first and second premolars, first molars at least).
* No previous orthodontic treatment.

Exclusion Criteria:

* Medically compromised patients.
* Patients suffering from any congenital or hereditary diseases.
* Smoking or any systemic diseases.
* Chronic use of any medications including antibiotics, phenytoin, cyclosporin, anti-inflammatory drugs, systemic corticosteroids, and calcium channel blockers.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Amount of intrusion | 6 months
  The amount the upper posterior teeth have been intruded.
Rate of bite closure | 6 months
  The rate by which the open bite closes as a result of posterior segment intrusion

SECONDARY OUTCOMES:
Average rate of intrusion | 6 months
  The amount of intrusion divided by the duration of intrusion
Root resorption | 6 months
  The amount of root resorption as a result of the intrusive force
Tipping | 6 months
  The amount of mesiodistal and buccolingual tipping of posterior teeth

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Participants data will not be exposed except for research committee